CLINICAL TRIAL: NCT01733147
Title: Modulation of Esophageal Inflammation in Barrett's Esophagus by Omega-3 Fatty Acids, a Double Blind Placebo Controlled Randomized Pilot Study
Brief Title: Modulation of Esophageal Inflammation in Barrett's Esophagus by Omega-3 Fatty Acids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Prasad G. Iyer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-005914
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Barrett's Esophagus; Obesity
Keywords: Omega-3 fatty acid
MeSH Terms: conditions — Barrett Esophagus; Obesity | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects with known Barrett's Esophagus (no dysplasia and low-grade dysplasia) will receive a placebo which looks exactly like the study drug, but contains no active ingredient, to be taken orally for six months.
  Interventions: Drug: Placebo
- Omega-3 polyunsaturated fatty acids (Active Comparator): Subjects with known Barrett's Esophagus (no dysplasia and low-grade dysplasia) will receive Omega-3 free fatty acids supplements to be taken orally for six months.
  Interventions: Drug: Omega-3 polyunsaturated fatty acids

INTERVENTIONS:
Drug: Omega-3 polyunsaturated fatty acids — 3 capsules a day of Omega 3 polyunsaturated fatty acids taken orally for six months; 2 capsules with breakfast and 1 capsule with their evening meal. Active drug will consist of 1200 mg of a ω3 FFA preparation containing 675 mg EPA and 300 mg DHA.
  Other Names: Docosahexaenoic Acid (DHA)/Eicosapentaenoic Acid (EPA)
  Arms: Omega-3 polyunsaturated fatty acids
Drug: Placebo — 3 capsules a day of placebo (1200 mg of ethyl oleate 3 capsules a day) taken orally for six months; 2 capsules with breakfast and 1 capsule with their evening meal.
  Arms: Placebo

SUMMARY:
This study is being done to understand the effect of dietary omega-3 fats in decreasing tissue inflammation in Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria

* Presence of BE defined as ≥ 1 cm of visible columnar mucosa in the distal esophagus with intestinal metaplasia on histology.
* Absence of high grade dysplasia or EAC on baseline histology.
* BMI > 30 kg/m2 or waist circumference > 102 cm in men, > 88 cm in women.
* Ability to give informed consent.

Exclusion Criteria

* Allergy to ω3 FFAs, fish or shellfish.
* Presence of high grade dysplasia or cancer on histology.
* Pregnant and or breastfeeding women
* Presence of esophagitis on initial endoscopy or symptoms of refractory GERD (heartburn or regurgitation ≥ 2 times a week) indicative of uncontrolled gastroesophageal reflux.
* Inability to give informed consent.
* Currently taking Omega3 FFA as prescription.
* Anti-coagulant therapy (Plavix, Warfarin, Coumadin)
* AST or ALT level > three times upper limit of normal at baseline
* LDL > 200 mg/dl at baseline.
* INR > 2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Iyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Omega-3 Polyunsaturated Fatty Acids
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omega-3 Polyunsaturated Fatty Acids | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58 to 73] | 66.5 [60 to 74] | 66 [60 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 25 | 19 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum PGE2 Levels
Description: Percent change from baseline to 6 months in serum prostaglandin E2 (PGE2) level obtained from blood draw
Time Frame: Baseline, 6 months
Measure: Median (Inter-Quartile Range); unit: Percentage of change in serum PGE2 level
Arm/Group | Placebo | Omega-3 Polyunsaturated Fatty Acids
Number analyzed (Participants) | 30 | 30
Percentage of change in serum PGE2 level | 4.44 [-33.20 to 59.06] | -21.65 [-59.64 to 5.07]

2. Primary Outcome: Change in Esophageal Tissue PGE2 Levels
Description: Percent change from baseline to 6 months in esophageal tissue prostaglandin E2 (PGE2) level obtained from endoscopic esophageal tissue collection
Time Frame: Baseline, 6 months
Measure: Median (Inter-Quartile Range); unit: Percentage of change in esophageal PGE2
Arm/Group | Placebo | Omega-3 Polyunsaturated Fatty Acids
Number analyzed (Participants) | 30 | 30
Percentage of change in esophageal PGE2 | 0.82 [-52.98 to 132.95] | 11.87 [-44.81 to 33.58]

3. Secondary Outcome: Change in Esophageal Macrophage Markers
Description: Percent change from baseline to 6 months in esophageal macrophage markers MCP-1 (Pro-inflammatory, M1 marker), CD 206 (Anti-inflammatory, M2 marker), and IL-10 (Anti-inflammatory, M2 marker) obtained from endoscopic esophageal tissue collection
Time Frame: Baseline, 6 months
Measure: Median (Inter-Quartile Range); unit: Percentage change in macrophage markers
Arm/Group | Placebo | Omega-3 Polyunsaturated Fatty Acids
Number analyzed (Participants) | 30 | 30
Percentage change in macrophage markers
  MCP-1 (Pro-inflammatory, M1 marker) | 4.81 [-0.27 to 12.47] | 2.12 [-4.8 to 17.25]
  CD 206 (Anti-inflammatory, M2 marker) | 4.19 [0.00 to 7.51] | 2.00 [-0.46 to 5.04]
  IL-10 (Anti-inflammatory M2 marker) | 1.91 [-0.87 to 3.27] | -0.53 [-3.25 to 1.06]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 6 months on all participants.
Arm/Group | Placebo | Omega-3 Polyunsaturated Fatty Acids
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | Omega-3 Polyunsaturated Fatty Acids (N=30)
Mild nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT01733147/Prot_SAP_000.pdf